CLINICAL TRIAL: NCT06692751
Title: The Value of Measuring Retinal Vascular Density by Optical Coherence Tomography-Angiography (OCT-A) in Patients with Microvascular Angina Confirmed by Myocardial Microcirculatory Resistance Index (MRI).
Acronym: EYE-NOCA
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: POMMIER J'InvEST-I 2023
Record Dates: First submitted 2024-11-15; First posted 2024-11-18 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-11

CONDITIONS: Microvascular Angina
MeSH Terms: conditions — Microvascular Angina | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- IMR<25: People without microvascular angina
  Interventions: Biological: Blood sampling; Procedure: Ophthalmological examination; Other: angina severity questionnaire
- IMR≥25: People with microvascular angina
  Interventions: Biological: Blood sampling; Procedure: Ophthalmological examination; Other: angina severity questionnaire

INTERVENTIONS:
Biological: Blood sampling — 2 tubes of 5 mL
Procedure: Ophthalmological examination — angiographic optical coherence tomography (OCT-A) on both eyes after pupil dilation.
  An optional 20-30 minute WLR may be offered following OCT-A.
Other: angina severity questionnaire — at inclusion, 3 months and 1 year Estimated filling time: 2 minutes

SUMMARY:
Microvascular angina is thought to affect around 112 million patients worldwide. However, this figure is underestimated due to the difficulty of making the diagnosis. It is a pathology caused by an alteration in the microcirculation of the heart muscle, which is not detectable on a standard coronary angiogram.

In view of its prognostic, therapeutic and medico-economic value, scientific societies currently recommend invasive measurement of the microcirculatory resistance index (MRI) to diagnose microvascular angina, in the absence of significant lesions on coronary angiography.

Several research teams, including our own, have shown that cardiovascular risk is associated with alterations in the vascularization of the small vessels (microcirculation) of the retina. Unlike the study of cardiac vessels, the study of retinal microcirculation using fundus photography (OCT-A) is simple, rapid, non-invasive and inexpensive. It appears to be an interesting alternative to the measurement of IMR for the diagnosis of microvascular angina.

This hypothesis has never yet been tested. The demonstration of an association between a decrease in retinal vascular density measured by OCT-A and an alteration in coronary microvascular function measured by IMR would pave the way for a completely non-invasive diagnosis of patients.

This is an observational, cohort, prospective, single-center pilot study comparing people who have received an IMR measurement as part of INOCA.

It is planned to include 158 participants. The overall follow-up period for each patient in the research is 12 months.

In routine care, IMR is measured during coronary angiography in patients presenting with ischemia on a non-invasive test and/or stress symptoms such as angina or dyspnea, for whom coronary angiography does not reveal any significant epicardial lesion.

Following this examination, two groups will be formed: a group with an IMR<25 and a group with an IMR≥25. Clinically, the study aims to determine the potential role of retinal OCT-A as a non-invasive examination for the diagnosis and/or follow-up of INOCA.

ELIGIBILITY:
Inclusion Criteria:

* Patients managed at Dijon University Hospital, having had an IMR measurement as part of INOCA during a coronary angiographic examination, consecutively includible, without angiographically or functionally significant coronary epicardial lesion (FFR < 0.80) explaining the clinical picture (= INOCA)
* Person having given oral consent
* Adult

Exclusion Criteria:

* Person not affiliated or not benefiting from a social security scheme
* Person subject to a legal protection measure (curatorship, guardianship) or a safeguard of justice measure
* Pregnant or breast-feeding women
* An adult incapable or unable to give consent
* Person with macular or retinal pathology, or severe bilateral myopia
* Person with genetic or idiopathic cardiomyopathy (dilated, hypertrophic or restrictive cardiomyopathy)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated at Dijon University Hospital, who received an IMR measurement as part of INOCA
Sampling Method: Non-Probability Sample
Enrollment: 158 (Estimated)
Dates: Start 2024-11-13 (Actual); Primary Completion 2027-11 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Retinal vascular density by "inner vessel length density" determined by OCT-A | At baseline

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Dijon Bourgogne, Dijon, France